CLINICAL TRIAL: NCT04613791
Title: Situation and Evolution of the Misuse of Alcohol and Other Addictive Behaviors in Obese Patients Being Managed at Nîmes University Hospital
Acronym: ADOB
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Other Study IDs: NIMAO/2019-2/FB-01
Record Dates: First submitted 2020-10-28; First posted 2020-11-03 (Actual); Last update posted 2023-01-12 (Actual); Status verified 2023-01

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity | interventions — Hematologic Tests; 4-amino-4'-hydroxylaminodiphenylsulfone; BES

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Two EDTA tubes of 5ml of blood will be collected for plasma extraction and conservation at -80°C in the biobank (samples taken at the same time as normal blood tests) .Samples will be stored in the hospital's bloodbank (biological resource centre) for the requirements of the future research programs or in view of giving them to other organisations for them to use for research. In order to be conformant with regulations, the samples collected will be subjected to a declaration and request for authorization with the authorities (Ministry of Further Education and Research and the Regional Health Agency) at the end of the trial.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Biological: Blood test — Collection of epidemio-clinical, biological, radiological and therapeutic patient data. Study samples collected from 154 patients to determine whether a particular immune profile could identify individuals prone to insulin resistance
  Other Names: Distribution of the following questionnaires: AUDIT, CAST, HADS, BES, Fagerstrom test and the EQVOD scale

SUMMARY:
Obesity is a multifactorial pathology in which external (lifestyle, environment) and internal (psychological or biological, especially genetic) factors are involved. These are responsible for a positive energy balance. One of the external factors that can intervene in the genesis of obesity is the existence of eating disorders: bulimic hyperphagia. Some teams consider bulimic hyperphagia as a form of addiction. After bariatric surgery, the appearance of new addictions has been observed.

In connection with Pr Perney's addictology department, the investigators have observed that some patients under treatment for obesity at the endocrinology department subsequently developed other addictions, in particular misuse of alcohol.

The hypotheses of this research are :

There appears to be a transfer from eating disorders to substance misuse addiction in post-treatment of obesity, particularly in patients who have undergone bariatric surgery.

The misuse of addictive substances most concerned by this transfer of addiction in the post-treatment of obesity, particularly after bariatric surgery, seems to be the misuse of alcohol.

This will be the first French cohort study on addictive behaviors in patients undergoing bariatric surgery and the first international study including non-operated obese patients benefiting from medical care alone. This study will improve the multidisciplinary management of these patients by integrating addictologists.

ELIGIBILITY:
* Patient being managed for the first time at Nîmes University Hospital Obesity Clinic ( complete hospitalization, outpatients' or consultation).
* Patient being managed for obesity defined by a body mass index (BMI) of 30 kg.m-² or over
* Patient affiliated to or covered by a health insurance scheme.
* Adult patient (≥ 18 years).

Exclusion Criteria:

* Patient with psychiatric disorder reducing capacity for comprehension.
* Patient in an exclusion period determined by another study.
* Patient under legal guardianship, tutorship or curatorship.
* Patient to whom it is impossible to give clear information
* Patient who is pregnant, about to give birth or breastfeeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The target population for this study corresponds to all patients being managed for obesity (Body Mass Index ≥ 30 kg.m-²).
  The source population for this study corresponds to all patients being managed by the obesity clinic at Nîmes University Hospital for obesity with a BMI ≥ 30 kg.m-² at the time of their first visit (complete hospitalization outpatients or consultation) for initiation to management (incident subjects).
Sampling Method: Non-Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2021-02-16 (Actual); Primary Completion 2023-12-15 (Estimated); Study Completion 2023-12-15 (Estimated)

PRIMARY OUTCOMES:
Presence of alcohol abuse evaluated at the first clinical consultation according to the AUDIT(Alcohol Use Disorders Identification Test) questionnaire. | Day 0
  The Alcohol Use Disorders Identification Test (AUDIT) self-questionnaire consists of 10 questions covering consumption (the first 3 questions), behaviors that may evoke dependency (not being able to stop drinking, inability to carry out one's plans, needing a drink in the morning) and problems related to alcohol consumption (guilt or remorse, memory loss, injuries, concerns from family and friends). Each question can be scored from 0 (low) - 4 (high) points, leading to a possible total score of 40 points. This questionnaire therefore makes it possible to cover all aspects of alcohol misuse in a very short space of time. It has been validated with good diagnostic performance: sensitivity at 92% and specificity at 94% for a threshold ≥ 8 (Saunders et al. 1993; Coulton et al. 2006). Moreover, this questionnaire is very widely used and recognized in scientific articles on addictology.
Presence of alcohol abuse evaluated at the first clinical consultation according to the AUDIT(Alcohol Use Disorders Identification Test) questionnaire. | Month 12
  The Alcohol Use Disorders Identification Test (AUDIT) self-questionnaire consists of 10 questions covering consumption (the first 3 questions), behaviors that may evoke dependency (not being able to stop drinking, inability to carry out one's plans, needing a drink in the morning) and problems related to alcohol consumption (guilt or remorse, memory loss, injuries, concerns from family and friends).Each question can be scored from 0 (low) - 4 (high) points, leading to a possible total score of 40 points. This questionnaire therefore makes it possible to cover all aspects of alcohol misuse in a very short space of time. It has been validated with good diagnostic performance: sensitivity at 92% and specificity at 94% for a threshold ≥ 8 (Saunders et al. 1993; Coulton et al. 2006). Moreover, this questionnaire is very widely used and recognized in scientific articles on addictology.
Presence of alcohol abuse evaluated at the first clinical consultation according to the AUDIT(Alcohol Use Disorders Identification Test) questionnaire. | Month 24
  The Alcohol Use Disorders Identification Test (AUDIT) self-questionnaire consists of 10 questions covering consumption (the first 3 questions), behaviors that may evoke dependency (not being able to stop drinking, inability to carry out one's plans, needing a drink in the morning) and problems related to alcohol consumption (guilt or remorse, memory loss, injuries, concerns from family and friends). Each question can be scored from 0 (low) - 4 (high) points, leading to a possible total score of 40 points.This questionnaire therefore makes it possible to cover all aspects of alcohol misuse in a very short space of time. It has been validated with good diagnostic performance: sensitivity at 92% and specificity at 94% for a threshold ≥ 8 (Saunders et al. 1993; Coulton et al. 2006). Moreover, this questionnaire is very widely used and recognized in scientific articles on addictology.
Presence of alcohol abuse evaluated at the first clinical consultation according to the DSM-5 questionnaire | Day 0
  The DSM-5 criteria are used to identify depression in all patients with high alcohol consumption (over14 glasses a week for women, 21 for men, or more than 4 glasses on one occasion). The DSM-5 outlines the following criterion to make a diagnosis of depression. The individual must be experiencing five or more symptoms during the same 2-week period and at least one of the symptoms should be either (1) depressed mood or (2) loss of interest or pleasure.
Presence of alcohol abuse evaluated at the first clinical consultation according to the DSM-5 questionnaire | Month 12
  The DSM-5 criteria are used to identify depression in all patients with high alcohol consumption (over14 glasses a week for women, 21 for men, or more than 4 glasses on one occasion). The DSM-5 outlines the following criterion to make a diagnosis of depression. The individual must be experiencing five or more symptoms during the same 2-week period and at least one of the symptoms should be either (1) depressed mood or (2) loss of interest or pleasure.
Presence of alcohol abuse evaluated at the first clinical consultation according to the DSM-5 questionnaire | Month 24
  The DSM-5 criteria are used to identify depression in all patients with high alcohol consumption (over14 glasses a week for women, 21 for men, or more than 4 glasses on one occasion). The DSM-5 outlines the following criterion to make a diagnosis of depression. The individual must be experiencing five or more symptoms during the same 2-week period and at least one of the symptoms should be either (1) depressed mood or (2) loss of interest or pleasure.

SECONDARY OUTCOMES:
Smoking (tobacco addiction) according to the Fagerström test | Day 0
  The Fagerström test consists of six questions. A score of 0 - 10 is obtained depending on the answers given. A score of 0 - 2 = zero addiction, 3 - 4 = slight addiction, 5 - 6 = moderate addiction, 7 ou 8 heavy addiction and 9 - 10 = very heavy addiction.
Smoking (tobacco addiction) according to the Fagerström test | Month 12
  The Fagerström test consists of six questions. A score of 0 - 10 is obtained depending on the answers given. A score of 0 - 2 = zero addiction, 3 - 4 = slight addiction, 5 - 6 = moderate addiction, 7 ou 8 heavy addiction and 9 - 10 = very heavy addiction.
Smoking (tobacco addiction) according to the Fagerström test | Month 24
  The Fagerström test consists of six questions. A score of 0 - 10 is obtained depending on the answers given. A score of 0 - 2 = zero addiction, 3 - 4 = slight addiction, 5 - 6 = moderate addiction, 7 ou 8 heavy addiction and 9 - 10 = very heavy addiction.
Cannabis addiction | Day 0
  The Cannabis Abuse Screening Test (CAST) questionnaire has 6 questions to which the answer YES (=1) or NO (=0) is given. A score ≥ 3 on the CAST indicates addiction to Cannabis.
Cannabis addiction | Month 12
  The Cannabis Abuse Screening Test (CAST) questionnaire has 6 questions to which the answer YES (=1) or NO (=0) is given. A score ≥ 3 on the CAST indicates addiction to Cannabis.
Cannabis addiction | Month 24
  The Cannabis Abuse Screening Test (CAST) questionnaire has 6 questions to which the answer YES (=1) or NO (=0) is given. A score ≥ 3 on the CAST indicates addiction to Cannabis.
Use of cocaine | Day 0
  The patient will be interviewed to find out whether he/she uses cocaine. This will be noted as Yes/No
Use of cocaine | Month 12
  The patient will be interviewed to find out whether he/she uses cocaine. This will be noted as Yes/No
Use of cocaine | Month 24
  The patient will be interviewed to find out whether he/she uses cocaine. This will be noted as Yes/No
Use of amphetamines | Day 0
  The patient will be interviewed to find out whether he/she uses amphetamines. This will be noted as Yes/No
Use of amphetamines | Month 12
  The patient will be interviewed to find out whether he/she uses amphetamines. This will be noted as Yes/No
Use of amphetamines | Month 24
  The patient will be interviewed to find out whether he/she uses amphetamines. This will be noted as Yes/No
Use of opioids | Day 0
  The patient will be interviewed to find out whether he/she uses opioids. This will be noted as Yes/No
Use of opioids | Month 12
  The patient will be interviewed to find out whether he/she uses opioids. This will be noted as Yes/No
Use of opioids | Month 24
  The patient will be interviewed to find out whether he/she uses opioids. This will be noted as Yes/No
Use of hallucinogenic drugs and/or new synthetic drugs | Day 0
  The patient will be interviewed to find out whether he/she uses hallucinogenic drugs and/or new synthetic drugs. This will be noted as Yes/No
Use of hallucinogenic drugs and/or new synthetic drugs | Month 12
  The patient will be interviewed to find out whether he/she uses hallucinogenic drugs and/or new synthetic drugs. This will be noted as Yes/No
Use of hallucinogenic drugs and/or new synthetic drugs | Month 24
  The patient will be interviewed to find out whether he/she uses hallucinogenic drugs and/or new synthetic drugs. This will be noted as Yes/No
Eating disorders | Day 0
  A score ≥ 17 on the BES (Binge Eating Scale) questionnaire indicates presence of an eating disorder.
Eating disorders | Month 12
  A score ≥ 17 on the BES (Binge Eating Scale) questionnaire indicates presence of an eating disorder.
Eating disorders | Month 24
  A score ≥ 17 on the BES (Binge Eating Scale) questionnaire indicates presence of an eating disorder.
Comorbidities | Day 0
  Presence of comorbidities for obesity (High blood pressure / Glucose intolerance or Diabetes / Sleep apnea syndrome / Dyslipidemia / Hepatic Steatosis / Cardiovascular diseases) will be noted from data in the patient file.
Comorbidities | Month 12
  Presence of comorbidities for obesity (High blood pressure / Glucose intolerance or Diabetes / Sleep apnea syndrome / Dyslipidemia / Hepatic Steatosis / Cardiovascular diseases) will be noted from data in the patient file.
Comorbidities | Month 24
  Presence of comorbidities for obesity (High blood pressure / Glucose intolerance or Diabetes / Sleep apnea syndrome / Dyslipidemia / Hepatic Steatosis / Cardiovascular diseases) will be noted from data in the patient file.
Quality of Life according to the EQVOD scale | Day 0
  The "Echelle de Qualité de Vie, Obésité et Diététique - EQVOD" (Quality of Life, Obesity and Dietetics Scale ) is a self-questionnaire validated in French which is adapted to the socio-cultural factors of obesity in France, making it possible to take into account the effects of dietary treatments on the quality of life of obese subjects (see Appendix 17.5) (Ziegler et al. 2005). It consists of 36 items, rated from 1 (always/highly) to 5 (never/not at all). It explores five dimensions (physical impact - Q1-Q11, psychosocial impact - Q12-Q22, impact on sexual life - Q23-Q26, food well-being - Q27-Q31 and diet experience - Q32-Q36). The rating for each dimension is reported as 100. The closer the score is to 100, the better the quality of life related to that dimension.
Quality of Life according to the EQVOD scale | Month 12
  The "Echelle de Qualité de Vie, Obésité et Diététique - EQVOD" (Quality of Life, Obesity and Dietetics Scale ) is a self-questionnaire validated in French which is adapted to the socio-cultural factors of obesity in France, making it possible to take into account the effects of dietary treatments on the quality of life of obese subjects (see Appendix 17.5) (Ziegler et al. 2005). It consists of 36 items, rated from 1 (always/highly) to 5 (never/not at all). It explores five dimensions (physical impact - Q1-Q11, psychosocial impact - Q12-Q22, impact on sexual life - Q23-Q26, food well-being - Q27-Q31 and diet experience - Q32-Q36). The rating for each dimension is reported as 100. The closer the score is to 100, the better the quality of life related to that dimension.
Quality of Life according to the EQVOD scale | Month 24
  The "Echelle de Qualité de Vie, Obésité et Diététique - EQVOD" (Quality of Life, Obesity and Dietetics Scale ) is a self-questionnaire validated in French which is adapted to the socio-cultural factors of obesity in France, making it possible to take into account the effects of dietary treatments on the quality of life of obese subjects (see Appendix 17.5) (Ziegler et al. 2005). It consists of 36 items, rated from 1 (always/highly) to 5 (never/not at all). It explores five dimensions (physical impact - Q1-Q11, psychosocial impact - Q12-Q22, impact on sexual life - Q23-Q26, food well-being - Q27-Q31 and diet experience - Q32-Q36). The rating for each dimension is reported as 100. The closer the score is to 100, the better the quality of life related to that dimension.
Anxiety and Depression | Day 0
  The Hospital Anxiety and Depression Scale (HADS) is a self-report questionnaire that assesses depressive and anxiety symptomatology (excluding somatic symptoms) and measures severity in patients between 16 and 65 years of age from a hospital environment (Zigmong & Snaith 1983, Snaith et al. 2003). The HADS consists of two parts: (a) 7 questions for screening for depression, and (b) 7 questions for screening for anxiety disorders. Each question receives a score between 0 and 3. The score for each part is obtained by adding the items that make up the part. The higher the score, the greater the severity of the corresponding symptoms.
  The French version was validated by Razavi et al. 1989 and Friedman et al. 2001.
Anxiety and Depression | Month 12
  The Hospital Anxiety and Depression Scale (HADS) is a self-report questionnaire that assesses depressive and anxiety symptomatology (excluding somatic symptoms) and measures severity in patients between 16 and 65 years of age from a hospital environment (Zigmong & Snaith 1983, Snaith et al. 2003). The HADS consists of two parts: (a) 7 questions for screening for depression, and (b) 7 questions for screening for anxiety disorders. Each question receives a score between 0 and 3. The score for each part is obtained by adding the items that make up the part. The higher the score, the greater the severity of the corresponding symptoms.
  The French version was validated by Razavi et al. 1989 and Friedman et al. 2001.
Anxiety and Depression | Month 24
  The Hospital Anxiety and Depression Scale (HADS) is a self-report questionnaire that assesses depressive and anxiety symptomatology (excluding somatic symptoms) and measures severity in patients between 16 and 65 years of age from a hospital environment (Zigmong & Snaith 1983, Snaith et al. 2003). The HADS consists of two parts: (a) 7 questions for screening for depression, and (b) 7 questions for screening for anxiety disorders. Each question receives a score between 0 and 3. The score for each part is obtained by adding the items that make up the part. The higher the score, the greater the severity of the corresponding symptoms.
  The French version was validated by Razavi et al. 1989 and Friedman et al. 2001.
Binge eating | Day 0
  The Binge Eating Scale (BES) is a self-administered questionnaire that diagnoses Binge Eating Disorder (BED) and assesses the behavioural, emotional and cognitive symptoms associated with Binge Eating Disorder in obese individuals (Gormally et al. 1982). It is composed of 16 items corresponding to groups of sentences including one to be selected from 3 to 4 propositions, which best describe how one feels. For each item, the subject has to choose the formulation that best corresponds to his current situation, which results in a score varying between 0 and 3 or between 0 and 2 for each item. Half of the items measure eating behaviours and the other half assess feelings or cognitions occurring during compulsive episodes. It gives a total score (from 0 to 46) that reflects the severity of the BED. A score greater than or equal to 18 indicates significant bulimic hyperphagia. The French version of this questionnaire was translated and validated by Brunault et al (2016).
Binge eating | Month 12
  The Binge Eating Scale (BES) is a self-administered questionnaire that diagnoses Binge Eating Disorder (BED) and assesses the behavioural, emotional and cognitive symptoms associated with Binge Eating Disorder in obese individuals (Gormally et al. 1982). It is composed of 16 items corresponding to groups of sentences including one to be selected from 3 to 4 propositions, which best describe how one feels. For each item, the subject has to choose the formulation that best corresponds to his current situation, which results in a score varying between 0 and 3 or between 0 and 2 for each item. Half of the items measure eating behaviours and the other half assess feelings or cognitions occurring during compulsive episodes. It gives a total score (from 0 to 46) that reflects the severity of the BED. A score greater than or equal to 18 indicates significant bulimic hyperphagia. The French version of this questionnaire was translated and validated by Brunault et al (2016).
Binge eating | Month 24
  The Binge Eating Scale (BES) is a self-administered questionnaire that diagnoses Binge Eating Disorder (BED) and assesses the behavioural, emotional and cognitive symptoms associated with Binge Eating Disorder in obese individuals (Gormally et al. 1982). It is composed of 16 items corresponding to groups of sentences including one to be selected from 3 to 4 propositions, which best describe how one feels. For each item, the subject has to choose the formulation that best corresponds to his current situation, which results in a score varying between 0 and 3 or between 0 and 2 for each item. Half of the items measure eating behaviours and the other half assess feelings or cognitions occurring during compulsive episodes. It gives a total score (from 0 to 46) that reflects the severity of the BED. A score greater than or equal to 18 indicates significant bulimic hyperphagia. The French version of this questionnaire was translated and validated by Brunault et al (2016).

OTHER OUTCOMES:
Age | Day 0
  Age will be recorded in years
Age | Month 12
  Age will be recorded in years
Age | Month 24
  Age will be recorded in years
Weight | Day 0
  Weight will be recorded in kg.
Weight | Month 12
  Weight will be recorded in kg.
Weight | Month 24
  Weight will be recorded in kg.
Height | Day 0
  Height will be recorded in cm
Height | Month 12
  Height will be recorded in cm
Height | Month 24
  Height will be recorded in cm
Sex | Day 0
  Male/Female
Sex | Month 12
  Male/Female
Sex | Month 24
  Male/Female
Other relevant items | Day 0
  All items (X-rays, biological tests, medicinal treatment…) relevant to the patient's care will be noted
Other relevant items | Month 12
  All items (X-rays, biological tests, medicinal treatment…) relevant to the patient's care will be noted
Other relevant items | Month 24
  All items (X-rays, biological tests, medicinal treatment…) relevant to the patient's care will be noted
Insulinemia only in the immun-Adob subpopulation | Day 0 and Month 12
  Method of determining insulin levels
Homa index in the Immun-Adob subpopulation | Day 0 and Month 12
  Blood glucose measurement that is routine test
Presence of waist circumference criterion ≥ 94 cm in men, ≥ 80 cm in women or BMI > 30 kg/m² | Day 0
  clinically determined visceral obesity
Triglyceride levels ≥ 1.5 G/L or treatment | Day 0
  Triglyceride measurements that are routine tests
Low HDL levels < 0.40g/L in men and < 0.50 in women or treatment | Day 0
  HDL measurement which is a routine biological analysis.
High blood pressure SBP ≥ 130 mmHg or DBP ≥ 85 mmHg or treatment. | Day 0
  Hypertension is determined clinically
Fasting blood glucose ≥ 1g/L | Day 0
  Glucose intolerance measurement which is a routine biological test.
Therelationship between membership in the immune activation profile of hyperinsulinism and the evolution of insulin levels | Between Day 0 and Month 12
  The percentages of CD57+, PD-1+, CD38+, HLA-DR+, naive or memory T4 or T8 cells will be determined by flow cytometry
The link between belonging to the immune activation profile of hyperinsulinism and the evolution of the HOMA index | Between Day 0 and Month 12
  The percentages of CD57+, PD-1+, CD38+, HLA-DR+, naive or memory T4 or T8 cells will be determined by flow cytometry
The link between the membership to the immune activation profile of hyperinsulinism and the evolution of the metabolic syndrome | Between Day 0 and Month 12

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Nimes, Nîmes, France